CLINICAL TRIAL: NCT07190664
Title: A Prospective, Randomized, Double-blind Study of Different Anesthesia Strategies for Postoperative Cough in Patients Undergoing Video-assisted Thoracoscopic Surgery
Brief Title: A Prospective, Randomized, Double-blind Study on the Effects of Different Anesthesia Strategies on Postoperative Cough in Patients Undergoing Video-assisted Thoracoscopic Surgery.
Acronym: Chronic cough
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025KY282
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Cough; Video-assisted Thoracoscopic Surgery (VATS)
Keywords: Video-assisted thoracoscopic surgery; chronic cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single-lumen endotracheal intubation group (Active Comparator): During the process of general anesthesia, a single-lumen endotracheal tube combined with a bronchial blocker was used to perform pulmonary isolation surgery, thereby meeting the requirements of video-assisted thoracoscopic partial lung resection.sample size:76
  Interventions: Other: Patients were randomly grouped
- Double-lumen endotracheal tube group (Active Comparator): During the general anesthesia process, a double-lumen endotracheal tube was used for lung isolation surgery, thus meeting the requirements of video-assisted thoracoscopic partial lung resection.sample size:76
  Interventions: Other: Patients were randomly grouped
- Laryngeal mask group (Experimental): During the general anesthesia procedure, a laryngeal mask was used, and the patient maintained spontaneous breathing for the thoracoscopic partial lung resection surgery.sample size:76
  Interventions: Other: Patients were randomly grouped

INTERVENTIONS:
Other: Patients were randomly grouped — All patients included in the study, were randomized

SUMMARY:
This study aims to systematically evaluate the effects of different anesthesia methods on postoperative chronic cough in lung cancer patients undergoing video-assisted thoracoscopic lung resection (VATS), and to clarify the effectiveness and safety of each anesthesia airway management strategy in reducing the incidence of postoperative chronic cough, shortening the duration of cough, alleviating the severity of symptoms, and improving the postoperative quality of life of patients.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, double-blind controlled study, aiming to explore the effects of different airway management strategies during surgery on the postoperative chronic cough in patients undergoing video-assisted thoracoscopic (VATS) lung resection. The study focuses on evaluating the incidence, duration, severity of postoperative chronic cough and its impact on patients' quality of life. It is expected to provide a basis for the prevention and intervention of postoperative chronic cough through prospective clinical data.

This study adopted a prospective, randomized, double-blind controlled design. The subjects were randomly divided into the single-lumen endotracheal tube group (Group A), the double-lumen endotracheal tube group (Group B), and the laryngeal mask airway group (Group C) in a 1:1:1 ratio to evaluate the effects of different airway management methods on postoperative chronic cough. The specific process is as follows: 1. Random sequence generation: The random grouping sequence was generated by independent non-clinical researchers using computer programs (such as SPSS, Excel or professional randomization tools), ensuring an equal distribution ratio, a repeatable process, and randomness. 2. Group information management: Each subject was assigned a unique random number, and this number and the group results were pre-loaded into opaque sealed envelopes and stored in order of the number. All envelopes were kept by a dedicated coordinator, who did not participate in the subsequent anesthesia or follow-up process to ensure the blinding of the grouping. 3. Group execution process: After the patient completed enrollment and signed the informed consent form, the research coordinator would open the envelope containing the subject's number before the operation, obtain the corresponding group information, and notify the anesthesiologist to execute the anesthesia strategy according to the predetermined grouping. The subjects and post-visit personnel remained blind to the grouping.

To ensure the ethical and safety aspects of the research, the following handling mechanisms have been established: 1. For patients who are not suitable for a certain anesthesia method before the operation: The anesthesiologist will conduct an assessment before the operation. If it is determined that they are not suitable for a certain anesthesia method, they will not proceed with the randomization process and will be registered as "Screening Failure", and will not be included in the intention-to-treat (ITT) analysis. 2. For those who need to change the intubation method due to uncontrollable factors during the operation (such as poor laryngeal mask ventilation and switching to intubation): Their original group will be retained for the ITT analysis. At the same time, a per-protocol (PP) analysis will be conducted in the data statistics for sensitivity analysis, and the reasons for the change will be detailed. 3. For those who did not complete the surgery during the operation or were lost to follow-up after the operation: If the subjects withdrew or were lost to follow-up, they will still be recorded as dropout and included in the dropout analysis. The endpoints to be included will be determined based on the degree of follow-up completion.

To reduce observation bias and analysis bias, this study was designed as a double-blind study. 1. Blind subjects: The postoperative visit personnel (responsible for assessing cough and quality of life scores) and data statisticians remained blind; the subjects were not clear about the intubation method during the operation (general anesthesia during the operation); the anesthesiologists were not blind (as they needed to perform the intubation operation). 2. Measures to ensure blinding: The anesthesiologists were not allowed to participate in any postoperative follow-up or data processing; the group information was hidden in the medical records and research forms, and was only identified by numbers.

The study observation period consists of two stages: the perioperative period and the postoperative chronic period. The follow-up time points during the perioperative period are on the 1st, 2nd, 3rd, 7th, 14th, and 1st month after the surgery; the follow-up time points during the postoperative chronic period are set at the 3rd, 6th, and 12th month after the surgery. The main focus of the study is to observe the incidence of postoperative chronic cough, the duration of coughing, the severity score, and the impact of coughing on quality of life. In addition, secondary indicators such as re-visits due to coughing and drug intervention can also be recorded to further evaluate the impact of the intervention measures on the long-term prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. planned wedge resection, segmentectomy or lobectomy;
2. more than 18 years old;
3. American Society of Anesthesiologists (ASA) grade ≤Ⅲ;
4. body mass index (BMI) ≤24 kg/m2;
5. Normal pulmonary function, predicted forced expiratory volume in 1 second (FEV1%) >50%, resting blood gas analysis showed arterial partial pressure of oxygen (PaO2) ≥75 mmHg and arterial partial pressure of carbon dioxide (PaCO2) <45 MMHG;
6. Normal cardiac function with ejection fraction (EF) > 50% of predicted value;
7. Informed consent and signed informed consent form.

Exclusion Criteria:

* (1) patients who refuse surgery and/or anesthesia; (2) preoperative pulmonary infection; (3) previous history of ipsilateral surgery or other medical history that may cause extensive pleural adhesions; (4) phrenic nerve palsy on the non-operative side; (5) patients with high risk of preoperative reflux (fasting <6 hours) or gastroesophageal reflux disease; (6) patients with heart, kidney, liver and other organ dysfunction and surgical contraindications; (7) with severe cognitive, psychological and communication disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative chronic cough, cough duration and cough severity score were recorded | The perioperative follow-up time points were 1 day, 2 days, 3 days, 7 days, 14 days and 1 month after operation. The follow-up time points of postoperative chronic phase were set at 3 months, 6 months and 12 months after operation.
  The perioperative follow-up time points were 1 day, 2 days, 3 days, 7 days, 14 days and 1 month after operation. The follow-up time points of postoperative chronic phase were set at 3 months, 6 months and 12 months after operation.